CLINICAL TRIAL: NCT01486836
Title: Evaluation of the Lumax DX ICD and the Linox DX Lead (ICD=Implantable Cardioverter Defibrillator, DX=Extended Diagnostics)
Brief Title: Lumax DX / Linox DX Evaluation
Status: Completed | Type: Observational
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Other Study IDs: 58
Record Dates: First submitted 2011-11-15; First posted 2011-12-07 (Estimated); Last update posted 2013-09-12 (Estimated); Status verified 2013-09

CONDITIONS: Cardiac Disease
Keywords: Cardiac disease (ICD indication)
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ICD therapy

SUMMARY:
The objective of this study is to investigate the safety and efficacy of the Lumax DX / Linox DX system.

No hypothesis has been defined.

ELIGIBILITY:
Inclusion Criteria:

* Patient meets the indication for ICD therapy
* LVEF ≥ 30%
* Patient's compliance with protocol
* Signed patient informed consent form

Exclusion Criteria:

* Patient meets one contraindication for ICD therapy
* Permanent atrial tachyarrhythmia
* Age < 18 years
* Cardiac surgery planned within the next 6 months
* Life expectancy of less than 6 months
* Limited contractual capability
* Participating in another clinical study of an investigational cardiac drug or device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with standard ICD indication who are referred to the hospital.
Sampling Method: Probability Sample
Enrollment: 38 (Estimated)
Dates: Start 2011-11; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Rate of appropriate atrial sensing | 3 months
Rate of successfully terminated tachyarrhythmia episodes | 3 months
Serious adverse device effect rate | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Charité Uniklinikum Benjamin Franklin, Berlin, Germany